CLINICAL TRIAL: NCT01583296
Title: Adaptation of a Behavioral Treatment for Latinos With Panic Disorder/Asthma
Brief Title: LUCHAR - Latinos Using Counseling for Help With Asthma and Anxiety Reduction
Acronym: LUCHAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Jonathan Feldman, Associate Professor of Psychology, Albert Einstein College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2009-223; R34MH087679 (NIH)
Record Dates: First submitted 2012-04-19; First posted 2012-04-24 (Estimated); Results first posted 2021-11-18 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-09

CONDITIONS: Asthma; Panic Disorder
MeSH Terms: conditions — Asthma; Panic Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CBT and HRVB (Experimental): Cognitive Behavioral Therapy (CBT) and Heart Rate Variability Biofeedback (HRVB)
  Interventions: Behavioral: CBT and HRVB
- Music Relaxation Therapy (MRT) (Active Comparator): Music Relaxation Therapy (MRT): music relaxation and breathing at resting respiration rate
  Interventions: Behavioral: Music Relaxation Therapy (MRT)

INTERVENTIONS:
Behavioral: Music Relaxation Therapy (MRT) — music relaxation therapy and breathing at resting respiration rate
  Arms: Music Relaxation Therapy (MRT)
Behavioral: CBT and HRVB — cognitive behavioral therapy and heart rate variability biofeedback
  Arms: CBT and HRVB

SUMMARY:
The research plan involves two aims: 1) Cultural adaptation of the Panic-Asthma Treatment and 2) a randomized, placebo-controlled pilot study. Participants will be primarily recruited from two major, inner-city hospitals in the Bronx, NY. Diagnosis of Panic Disorder (PD) will be based on the Structured Clinical Interview for DSM-IV. Diagnosis of asthma will be based on national guidelines. The first year of the project will be devoted to approximately 5 focus groups with Latino (primarily Puerto Rican) participants, pilot treatment and participant feedback. The protocol will be adapted based on key cultural issues that are systematically observed during Phase 1. During Years 2-3, 40 participants with PD and asthma will be randomized into two treatment arms: Panic-Asthma Treatment and an active placebo condition involving music therapy and paced breathing at resting respiration rates. Each treatment will involve 8 weekly sessions. An interviewer, who will be blind to treatment condition, will conduct assessments at pre-treatment, mid-treatment, post-treatment, and 3-month follow-up. The primary hypotheses are that participants in the Panic-Asthma treatment group will have greater decreases than subjects in the placebo condition on the PD severity scale and albuterol use (i.e., rescue asthma medication) from pre-test to post-test and across 3-month follow-up.

DETAILED DESCRIPTION:
Asthma and panic disorder (PD) share strikingly similar phenomenology. Respiratory related symptoms, such as dyspnea, dizziness, chest tightness, feelings of choking and sensations of smothering are common in both disorders. The overlap in symptoms between asthma and panic may lead an individual to mistake a panic attack as an asthma attack. In order to better understand this overlap, we hypothesized that participants who received Cognitive Behavioral Psychophysiological Therapy (CBPT) would display greater reductions in PD severity and improvements in asthma control at post- treatment and 3-month follow-up. We predicted that improvements in PD severity in the CBPT group would be mediated by reductions in the perceived physical consequences of anxiety. We selected music therapy and paced breathing at each participant's average respiration rate for the comparison active treatment. Randomized participants will undergo either the CBPT or MRT protocol, be given the same psychological assessments, and have their physiological data collected.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV criteria for current PD with or without agoraphobia
* fluency in spoken English or Spanish
* no changes in prescribed levels of panicolytic medication for two months prior to the study and no changes in panicolytic medication during the two months of the active protocol
* history or presence of episodic symptoms of airflow obstruction, namely, wheezing, shortness of breath, chest tightness, or cough
* airflow obstruction showing FEV1 < 80% predicted and FEV1/FVC < 65% or below the lower limit of normal
* airflow obstruction must be at least partly reversible, as demonstrated by:
* Positive Bronchodilator test in past year from Medical Chart Review or Baseline session
* Positive Bronchodilator test during past 10 years (from Medical Chart Review) and asthma symptoms reported past 12 months (from Medical Chart Review or Baseline Questionnaires)
* Improvement in PEF of ≥20% from Medical Chart Review past 10 years (from Medical Chart Review) and asthma symptoms reported past 12 months (from Medical Chart Review or Baseline Questionnaires)
* Clinical improvement in asthma symptoms after initiation of anti-inflammatory medication, as documented in medical records.

Exclusion Criteria:

* evidence of active bipolar disorder or psychosis
* mental retardation or organic brain syndrome
* current alcohol or substance abuse/dependence
* foreign body aspiration, vocal cord dysfunction, or other pulmonary diseases
* history of smoking 20 pack-years or more
* history consistent with emphysema, sarcoidosis, bronchiectasis, pulmonary tuberculosis, lung cancer, cardiovascular or neurological disease
* current participation in alternative psychotherapy for anxiety or panic for less than 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2010-07; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Feldman, PhD, Principal Investigator — Albert Einstein College of Medicine
Locations (2):
- United States (2):
  - Jacobi Medical Center/North Central Bronx Hospital (NBHN), The Bronx, New York
  - Montefiore Medical Center: Moses Division/Weiler Division, The Bronx, New York

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CBT and HRVB | Music Relaxation Therapy (MRT)
Started | 27 | 26
Completed | 16 | 16
Not Completed | 11 | 10
Not completed — Withdrawal by Subject | 11 | 10

BASELINE CHARACTERISTICS:
Population: While 27 participants were allocated to the CBPT intervention, 3 dropped out before the baseline session. Similarly, 26 participants were allocated to the MRT intervention but 2 dropped out before the baseline session. Accordingly, in each of the study arms 24 participants completed the baseline session.
Groups:
- Total: Total of all reporting groups
Arm/Group | CBT and HRVB | Music Relaxation Therapy (MRT) | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.8 (11.8) | 42.6 (12.9) | 43.2 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 23 | 45
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24 | 24 | 48
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States: Continental US-Born | 14 | 13 | 27
  United States: Non-Continental US-Born | 10 | 11 | 21
Household Income [Count of Participants; unit: Participants]
  >$16000 | 10 | 14 | 24
  < $16000 | 14 | 10 | 24
Education [Count of Participants; unit: Participants]
  At least some college | 8 | 14 | 22
  High School | 6 | 7 | 13
  Less than high school | 10 | 3 | 13
Marital Status [Count of Participants; unit: Participants]
  Married | 6 | 5 | 11
  Never married | 11 | 11 | 22
  Separated/Divorced/Widowed | 7 | 8 | 15
Employment Status [Count of Participants; unit: Participants]
  Employed or Student | 9 | 9 | 18
  Unemployed | 15 | 15 | 30
Health Insurance [Count of Participants; unit: Participants]
  Medicaid or Medicare | 21 | 20 | 41
  Other | 3 | 4 | 7
Cigarette Smoking History [Count of Participants; unit: Participants]
  Current Smoker | 5 | 6 | 11
  Ex-Smoker | 6 | 3 | 9
  Never Smoked | 13 | 15 | 28
Asthma Severity [Count of Participants; unit: Participants]
  Intermittent/Mild Persistent | 3 | 4 | 7
  Moderate Persistent | 19 | 19 | 38
  Severe Persistent | 2 | 1 | 3
Language [Count of Participants; unit: Participants]
  English | 20 | 17 | 37
  Spanish | 4 | 7 | 11

OUTCOME MEASURES:

1. Primary Outcome: Change in Severity of Panic Disorder as Measured by the Panic Disorder Severity Scale
Description: The Panic Disorder Severity Scale (PDSS) is a clinician-administered questionnaire used to assess the severity of panic attacks. The PDSS consists of seven items with each ranging in severity from 0 (none) - 4 (extreme); so total score ranges from 0 to 28.
Time Frame: Baseline, Post-Treatment (end of week 8)
Population: While 27 participants were allocated to the CBPT intervention, 3 dropped out before the baseline session. Similarly, 26 participants were allocated to the MRT intervention but 2 dropped out before the baseline session. Accordingly, outcome measures were analyzed for the 48 participants (24 in each arm) that completed their baseline sessions.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CBT and HRVB | Music Relaxation Therapy (MRT)
Number analyzed (Participants) | 24 | 24
score on a scale
  Baseline | 2.17 (0.16) | 2.40 (0.17)
  Post-Treatment | 1.64 (0.18) | 1.52 (0.19)

2. Primary Outcome: Asthma Control Based on Rescue Medication Use
Description: Dosers (electronic devices used to monitor the usage of metered-dose inhalers) were attached to participants' asthma rescue inhalers to count the number of puffs of medication used during the treatment period. Use of rescue medication was then coded as good asthma control (less than or equal to rescue medication use twice a week) or poor control (rescue medication use greater than two days a week) in accordance with national guidelines (NHLBI, 2007).
Time Frame: Change from Baseline to Post-Intervention (8 weeks)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: % good asthma control
Arm/Group | CBT and HRVB | Music Relaxation Therapy (MRT)
Number analyzed (Participants) | 24 | 24
% good asthma control
  Baseline | 28.99 (10.69) | 23.24 (9.69)
  Post-Treatment | 55.42 (12.83) | 51.48 (13.36)

3. Primary Outcome: Clinical Global Impression Scale (CGI)
Description: The CGI is a 2-item scale rated by clinicians to assesses for a patient's functioning prior and subsequent to the implementation of an intervention. In the current study, the CGI was used to assess panic disorder illness severity in patients as well as identify whether subjects responded to the study intervention. The CGI scale includes a question on level of improvement subsequent to intervention ranging from 1 (very much improved) to 7 (very much worse), and a question on severity of illness ranging from 1 (normal) to 6 (among the most extremely ill of patients). To be a treatment responder, a participant had to have a score of 2 (much improved) or better and be rated as a 3 (mild) or less on their illness severity.
Time Frame: Change from Baseline to Post-Intervention (8 weeks)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | CBT and HRVB | Music Relaxation Therapy (MRT)
Number analyzed (Participants) | 24 | 24
Participants
  Responders | 7 | 5
  Non-Responders | 17 | 19

4. Secondary Outcome: Asthma Control Questionnaire (ACQ)
Description: The ACQ is a self-report questionnaire to assess asthma control based on asthma symptoms, nighttime awakenings, and use of rescue medication for asthma. Each item is given a score from 0 to 6 with lower scores indicating better asthma control. The ACQ total scale score is an average of the item questions, with scores ranging between 0 (well controlled) and 6 (extremely poorly controlled).
Time Frame: Change from Baseline to Post-Intervention (8 weeks)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: natural log transformed score on a scale
Arm/Group | CBT and HRVB | Music Relaxation Therapy (MRT)
Number analyzed (Participants) | 24 | 24
natural log transformed score on a scale
  Baseline | 0.85 (0.14) | 0.85 (0.15)
  Post-Treatment | 0.22 (0.17) | 0.46 (0.18)

5. Secondary Outcome: Medication Adherence Report Scale (Adherence to Controller Medications for Asthma)
Description: Self-report measure of adherence to controller medications with 10 items ranging from 1 (always) to 5 (never). Higher mean scores indicate greater adherence and a score > 4.5 is considered good adherence.
Time Frame: Change from Baseline to Post-Intervention (8 weeks)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CBT and HRVB | Music Relaxation Therapy (MRT)
Number analyzed (Participants) | 24 | 24
score on a scale
  Baseline | 3.51 (0.17) | 4.38 (0.18)
  Post-Treatment | 4.15 (0.17) | 4.40 (0.20)

ADVERSE EVENTS:
Time Frame: Data on participant adverse events were collected over the course of approximately 3 months, from the participant's baseline session to their 3- month follow-up session.
Description: The study utilized the clinicaltrials.gov definition of adverse events. At each study session participants were asked if any adverse events had occurred since the last study session, with the PI reporting any deaths and serious events (within 48 hours of PI's knowledge) and Unanticipated Events (within 30 days of PI's knowledge) to the IRB committee.
Arm/Group | CBT and HRVB | Music Relaxation Therapy (MRT)
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24

LIMITATIONS AND CAVEATS:
The main limitations of this study were the small sample size and high drop-out rate (40%). The MARS was not applicable to 25% of participants who were not taking ICS medications. The use of %FEV1 as the sole measure of pulmonary function was limited by its snapshot measure of asthma control. Finally, the findings of this study are specific to a narrow sample of Latinos and may not generalize.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No